CLINICAL TRIAL: NCT00914355
Title: Phase II Trial of Stereotactic Body Radiation Therapy for Unresectable Hepatocellular Carcinoma
Brief Title: Stereotactic Body Radiation Therapy (SBRT) Hepatocellular Carcinoma (COLD 2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 07-0346-C
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Stereotactic Body Radiation; Unresectable liver cancer; Patients with Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SBRT for Hepatocellular Carcinoma (Experimental)
  Interventions: Radiation: Stereotactic Body Radiation

INTERVENTIONS:
Radiation: Stereotactic Body Radiation — Radiation therapy will be delivered on six occasions, over two weeks. Each treatment will take approximately 30 minutes to deliver.You may be asked to swallow 250 cc of oral contrast before each radiation therapy treatment.Pepto Bismol (a liquid that coats the stomach and is used to treat heartburn) and/or water may be combined with the contrast to improve the quality of the stomach's image.

SUMMARY:
This study is designed to see whether stereotactic body radiation therapy (SBRT) can reduce tumour size, slow progression of the disease, prolong life and improve quality of life of patients with hepatocellular carcinoma, a cancer of the liver, that cannot be removed surgically (unresectable) and cannot be treated with ablative therapy (e.g. radio-frequency ablation) or trans-arterial chemo-embolization (TACE) therapy (delivery of chemotherapy through an artery that feeds into the liver). SBRT is concentrated focused radiation therapy delivered very precisely to the liver tumour. It is hoped that knowledge obtained from this study will improve our ability to treat patients with liver tumours that cannot be treated with surgery and other methods, and that SBRT may prove to be a treatment that can lead to long-term and permanent control of liver tumours for some patients.

DETAILED DESCRIPTION:
From July 2003 to May 2007, over 40 patients with hepatocellular carcinoma participated in two studies at Princess Margaret Hospital (PMH) designed to determine the safety of treating hepatocellular carcinoma with SBRT. These studies have shown that SBRT can be delivered safely to the majority of patients with hepatocellular carcinoma. The treated tumour was controlled (shrank or remained the same size) in 78% of patients at one year following treatment.The median survival of patients was 11 months (i.e. half of patients survived longer and half shorter than 11 months). This survival rate is better than that expected in patients treated with supportive care only (no treatment other than care to make you feel better). Supportive care patients have a median survival rate of 3-9 months. We expect that the benefits of SBRT in this study will be similar to those observed in our initial studies.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pathologically, 2)diagnosed by showing vascular enhancement of the lesion on at least two imaging techniques, or 3) diagnosed by showing vascular enhancement on a single technique if the AFP is greater than 200, in the setting of cirrhosis or chronic hepatitis B without cirrhosis (EASL consensus conference guidelines).
* Either 1) the tumour must be unresectable, based on the opinion of an experienced surgeon specializing in hepatic resection, or 2) the patient Phase II SBRT HCC 13 must be medically inoperable, or 3) extra-hepatic metastases must be present (making hepatic surgery an inappropriate treatment option).
* Karnofsky performance status (KPS) > 60 (Appendix II)
* Age: 18 years or older. Both male & female patients of all races can be included in this study. Female patients within reproductive years may not be, nor become, pregnant during participation in this study
* Patients must have recovered from the effects of previous therapy.
* Maximal tumor size of 15 cm.
* Adequate organ function as assessed as follows:

  * Hemoglobin > 90 g/L
  * Absolute neutrophil count > 1.0 bil/L
  * Platelets > 50 bil/L
  * Bilirubin < 4.0 times upper range of normal
  * INR < 1.5 or correctable with vitamin K (unless patient is on coumadin in which case higher levels are acceptable)
  * AST or ALT < 6.0 times upper range of normal
* Child's A 5-6 liver score or Child B 7-8 liver score, which is only permitted if the maximal tumor size is 10 cm
* Previous liver resection or ablative therapy is permitted.
* Life expectancy > 3 months
* The volume of uninvolved must be at least 700 cc
* Up to five discrete liver tumors
* Patients must have signed a study-specific informed consent form. If the patient's mental status precludes this, written informed consent may be given by the patient's legal representative.

Exclusion Criteria:

* Patients with active hepatitis or encephalopathy related to liver failure
* Prior radiation therapy to the right upper abdomen, precluding reirradiation of the liver. That is, any previous radiation therapy in which a mean dose to the liver of 15 Gy in conventional fractionation was delivered, or previous doses to critical normal structures that would make re-irradiation unsafe. The PI should be called if there is any question of safety of re-irradiation.
* Eligible for RFA or alcohol ablation
* Eligible for TACE
* Prior uncontrolled, life threatening malignancy within the six months.
* Pregnancy is not permitted, and in women of child bearing age, a pregnancy test and acceptable methods of contraception are warranted.
* Previous gastric, duodenal or variceal bleed within the past 2 months.
* Commencement of coumadin use within the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-08; Primary Completion 2020-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Determine one year local progression free rate, defined as lack of progression within the irradiated volume, using RECIST criteria | 5 years

SECONDARY OUTCOMES:
Overall progression free survival | 5 years
Overall survival | 5 years
Quality of life | 5 years
CTC3.0 toxicity | 5 years
Cytokine response to radiation and association with complications | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dawson, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Bujold A, Massey CA, Kim JJ, Brierley J, Cho C, Wong RK, Dinniwell RE, Kassam Z, Ringash J, Cummings B, Sykes J, Sherman M, Knox JJ, Dawson LA. Sequential phase I and II trials of stereotactic body radiotherapy for locally advanced hepatocellular carcinoma. J Clin Oncol. 2013 May 1;31(13):1631-9. doi: 10.1200/JCO.2012.44.1659. Epub 2013 Apr 1. PMID 23547075